CLINICAL TRIAL: NCT02427932
Title: PK and PD Modeling of Ampicillin and Gentamicin in Peripartum Patients
Brief Title: Pharmacokinetic (PK) and Pharmacodynamic (PD) Modeling of Ampicillin and Gentamicin in Peripartum Patients
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: David Drover, MD (Unknown)
Responsible Party: Principal Investigator, Brendan Carvalho, MBBCh, FRCA, MDCH, Associate Professor, Dept. of Anesthesia, Stanford University
Other Study IDs: 29664
Record Dates: First submitted 2015-04-14; First posted 2015-04-28 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Drug Metabolism During Pregnancy
Keywords: Pharmacokinetics (PK); Pharmacodynamics (PD)
MeSH Terms: interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pregnant/Ampicillin: pregnant participants who will receive Ampicillin for conditions such as Group B Streptococcus
  Interventions: Drug: Ampicillin
- Non-pregnant/Ampicillin: non-pregnant participants who will receive Ampicillin for a qualifying hospital admission
  Interventions: Drug: Ampicillin
- Pregnant and Non-pregnant/Ampicillin and Gentamicin: pregnant participants who will receive Ampicillin and Gentamicin for conditions such as chorioamnionitis; non-pregnant participants who will receive Ampicillin and Gentamicin for a qualifying hospital admission
  Interventions: Drug: Ampicillin and Gentamicin
- Non-Pregnant/Gentamicin: non-pregnant participants who will receive Gentamicin for a qualifying hospital admission
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Ampicillin — Pregnant participants will receive Ampicillin 2g IV loading dose followed by 1g IV every 4 hrs until delivery for Group B Strep prophylaxis; non-pregnant participants will receive Ampicillin for qualifying diagnosis
  Groups: Non-pregnant/Ampicillin; Pregnant/Ampicillin
Drug: Ampicillin and Gentamicin — Pregnant participants will receive Ampicillin 2g IV every 6hrs along with Gentamicin 5mg/kg IV every 24 hrs for chorioamnionitis; non-pregnant participants will receive for qualifying diagnosis
  Groups: Pregnant and Non-pregnant/Ampicillin and Gentamicin
Drug: Gentamicin — Prescribed to non-pregnant participants
  Groups: Non-Pregnant/Gentamicin

SUMMARY:
This study proposes to compare the metabolism of Ampicillin and Gentamicin by pregnant women to that of non-pregnant women; the placental transfer over time; and the subsequent metabolism of the transferred drug(s) in the neonate.

DETAILED DESCRIPTION:
Pregnant women who present to Labor and Delivery will be identified as potential participants based on Inclusion/Exclusion criteria and their need to receive Ampicillin and/or Gentamicin therapy. The additional group of 20 non-pregnant women will also be identified based on Inclusion/Exclusion criteria and their need to receive Ampicillin and/or Gentamicin therapy.

Once identified, interested candidates will be fully informed of the study procedures, have all questions answered, and informed consent obtained.

Pregnant participants will receive Ampicillin 2g IV loading dose followed by 1g IV every 4 hrs until delivery; or Ampicillin 2g IV every 6hrs along with Gentamicin 5mg/kg IV every 24 hrs. Dose times will be recorded.

Non-pregnant participants will receive similar doses of either Ampicillin and/or Gentamicin, if not the same dose(s).

Fingerstick blood collection will be drawn from both populations at the following timepoints:

* before the administration of Ampicillin, and/or
* before the administration of Gentamicin
* after the full initial dose of the antibiotic has infused, at 5 min, 15 min, 30 min, 2-3hr, 4-6hr, immediately prior to the next dose of drug, and at DELIVERY (a 5 minute window for each timepoint will be permitted) If delivery occurs prior to the 3 or 6 hr timepoints, fingerstick blood collection should continue

Samples will be obtained on filter paper via the Dry Blood Spot (DBS) method, which is clinically appropriate for the purposes of this study.

Umbilical venous and arterial blood will also be drawn for sampling from the placenta after delivery, and cutting of the umbilical cord.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, pregnant woman (28-42 weeks)
* Generally healthy, non-pregnant female
* Scheduled to receive Ampicillin and/or Gentamicin IV
* Ages 18-55 years old
* Relatively normal Comprehensive Metabolic Panel (if available), as evidenced by recent blood work
* Able and willing to sign consent

Exclusion Criteria:

* Women with known renal or hepatic impairment; preeclampsia; Diabetes, including Gestational; any medical condition that, in the opinion of the Investigator or research team member, could potentially interfere with the study objectives
* Women who are participating in another study
* Pregnant with multiples
* BMI > 40

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women receiving ampicillin or gentamicin
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profiling to Measure Maternal Metabolism of Ampicillin and/or Gentamicin in Pregnancy | predose; after the full initial dose of the antibiotic has infused, at 5min, 15min, 30min, 2-3hr, 4-6hr, immediately prior to the next dose of drug, and at DELIVERY
  blood samples will be taken at the above timepoints; data analysis of all specimens will begin approx. 12-15 months from start of study

SECONDARY OUTCOMES:
Profile of Neonatal Metabolism of Ampicillin and Gentamicin That Crosses the Placental Barrier | At delivery/upon cutting of umbilical cord
  blood samples to be drawn at the above timepoint; data analysis of all specimens will begin approx. 12-15 months from start of study
PD Modeling of Peripartum Patients Receiving Ampicillin and/or Gentamicin | predose; while dosing; post dose
  subject will be observed for adverse events related to drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh, Study Director — Stanford University; David Drover, MD, Study Director — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States